CLINICAL TRIAL: NCT04981262
Title: Improved Quality of Life in Children With Intestinal Failure - a Randomised Intervention Trial
Brief Title: Improved Quality of Life in Children With Intestinal Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Rut Anne Thomassen, Clinical Dietitian, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170851
Record Dates: First submitted 2021-06-22; First posted 2021-07-28 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Intestinal Pseudo-Obstruction; Short Bowel Syndrome; Malabsorption Syndrome Autoimmune Enteropathy; Bacterial Overgrowth
MeSH Terms: conditions — Intestinal Pseudo-Obstruction; Short Bowel Syndrome; Autoimmune enteropathy

STUDY DESIGN:
Intervention Model Description: Intervention with prebiotics to all participants for 4 weeks. Then randomisation to continue with prebiotics for 6 months or no intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stimulance (Experimental): 4 weeks intervention with Stimulance for all participants
  Interventions: Dietary Supplement: Stimulance
- Stimulance 6 months (Experimental): 6 months intervention
  Interventions: Dietary Supplement: Stimulance
- No intervention (No Intervention): 6 months control group

INTERVENTIONS:
Dietary Supplement: Stimulance — Intervention with Prebiotic supplement
  Arms: Stimulance; Stimulance 6 months

SUMMARY:
Children with intestinal failure have a lack of tolerance for food in the intestine. The children are dependent on intravenous nutrition over a long period of time period to ensure growth and development. The condition is characterized by bacterial overgrowth in the intestine, with nausea, vomiting, diarrhea and flatulence as physical symptoms. Mental health is affected in the form of lower quality of life, lack of school participation and less social contact with peers. The investigators own (unpublished) data show that children with intestinal failure have a lower quality of life than healthy people. Standard treatment is antibiotics, but the effect of these is short-lived, and many must have repeated courses. Prebiotics are indigestible carbohydrates (fiber) in foods that positively affect the bacterial flora and promote intestinal health. In this project the investigators want to see if supply of prebiotics can change the bacterial balance, reduce symptoms of bacterial overgrowth and increase quality of life. The study is unique, as Prebiotics have not previously been used in the treatment of intestinal failure. If successful, it can pave the way for a new and better treatment method that can potentially be transferred to other conditions with imbalance in the intestinal flora. The study is a randomized intervention study and is consist of two phases. In phase 1, the effect of 4 weeks of open intervention with prebiotics is studied to establish so-called "proof of concept". Data from phase 1 are used to look at connections between the composition of intestinal flora, nutritional status and bowel function. The intervention involves the use of a prebiotic product (Stimulance, Nutricia), which is added to childs regular food. In phase 2, patients are randomized into two groups. One group will continue with the product for 6 months, while the other group does not receive prebiotics.

DETAILED DESCRIPTION:
Quality of life, gastrointestinal symptoms and family impact are measured using validated forms for four weeks before intervention phase 1, at start-up and after phase 1, as well as after phase 2. Stool samples are collected at the same time points. Weight, height is measured and blood tests are collected at the start and end of phases 1 and 2. Data on diet and nutritional treatment are collected at the start and end of the two phases. The stool samples are analyzed for short fatty acids (marker for good intestinal health), the composition of the intestinal flora and inflammation markers. Blood samples are analyzed for infection markers, intestinal health markers and nutritional markers. Nutritional data are analyzed for nutrient content and the dependence on nutritional support is calculated.

The investigators expect that the study will lead to an improved quality of life for the patient group through increased tolerance to food in the intestine, reduced antibiotic use and reduction of gastrointestinal symptoms. The project is patient-oriented.

ELIGIBILITY:
Inclusion criteria are:

* Diagnosed with congenital malformations or diseases requiring intestinal surgery leading to short bowel syndrome or
* Diagnosed with conditions and diseases leading to intestinal failure e.g pseudo obstruction.

And Treated with parenteral nutrition for minimum 60 days within a 74 day period.

Exclusion criteria:

* Children in need of temporary advanced nutrition intervention due to illness, e.g. infections.
* Children with temporary malfunctioning gut due to advanced medical treatment, for example cancer treatment or transplantation

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-12-02 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in Quality of life scores before and after treatment with prebiotics | 6 months
  Changes in Pediatric quality of life inventory scores on an analog scale from 0-100 where higher scores means better outcome
Changes in gastro intestinal symptoms scores before and after treatment with prebiotics | 6 months
  Pediatric quality of life inventory Gastro intestinal symptom scale scores on an analog scale from 0-100 where higher scores means better outcome
Changes in familt impact scores before and after treatment with prebiotics | 6 months
  Pediatric quality of life inventory Family Impact Module scores on an analog scale from 0-100 where higher scores means better outcome

SECONDARY OUTCOMES:
Changes in Microbiota | 6 months
  Measured by Short Chain Fatty Acids and microbiota composition

CONTACTS AND LOCATIONS:
Overall Officials: Rut Anne Thomassen, Principal Investigator — Oslo University Hospital; Anne Charlotte Brun, MD PhD, Study Director — Oslo University Hospital; Christine Henriksen, PhD, Study Chair — University of Oslo
Locations (1):
- Oslo University Hopspital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomassen RA, Kvammen JA, Bentsen BS, Bratlie M, Bohn SK, Farstad H, Kahrs C, Ngo L, Nybo C, Saeland C, Tjora E, Tronstad RR, Stordal K, Brun AC, Henriksen C. Effect of prebiotics on gastrointestinal symptoms and quality of life in children with intestinal failure: A pilot study. J Pediatr Gastroenterol Nutr. 2025 Oct;81(4):975-985. doi: 10.1002/jpn3.70186. Epub 2025 Aug 6. PMID 40770855

DOCUMENTS (1):
  • Study Protocol (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT04981262/Prot_000.pdf